CLINICAL TRIAL: NCT06159296
Title: Randomised, Placebo-controlled, Double-blind Cross-over Study to Investigate the Therapeutic Effects of an Inhaled Hydrogen/Oxygen Mixture to Improve Long COVID Symptoms
Brief Title: Effect of Inhaled Hydroxy Gas on Long COVID Symptoms
Acronym: LCHydroxy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr. Shakeeb H Moosavi, Reader in Clinical Physiology, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 231692
Record Dates: First submitted 2023-12-02; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Post-Acute COVID-19 Syndrome; Long COVID; Long Haul COVID-19; Long-Haul COVID; Post-Acute Sequelae of COVID Infection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned a machine that delivers either hydroxy or placebo gas in the first three weeks of the study. Those who receive placebo in the first three weeks will receive hydroxy in the last three weeks following a minimum of a 3 week washout period. Those who receive hydroxy in the first three weeks will receive placebo in the last three weeks.
Who Masked: Participant, Investigator
Masking Description: The study is double blind. The participants will not know whether the machine they use delivers hydroxy or placebo gas. The PI and outcome assessors will also not know which machine delivers hydroxy or placebo gas to participants during the running of the study. A collaborator will be in charge of blinding for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-Placebo arm (Other): The participants in this arm are given a machine that produces hydroxy gas in the first three weeks. In the final three weeks of the study, they will use a machine that produces a placebo gas.
  Interventions: Device: Hydroxy gas
- Placebo-treatment arm (Other): The participants in this arm are given a machine that produces a placebo gas in the first three weeks. In the final three weeks of the study, they will use a machine that produces hydroxy gas.
  Interventions: Device: Hydroxy gas

INTERVENTIONS:
Device: Hydroxy gas — Hydroxy gas is a combination of hydrogen and oxygen together.

SUMMARY:
The goal of this clinical trial is to see if several weeks of self-administered, home-based, treatment involving breathing hydroxy gas (a mixture of hydrogen and oxygen) for at least 2 hours a day for 3 weeks, will relieve symptoms in patients suffering from Long COVID. The main question it aims to answer is whether inhaling hydroxy gas might be a useful treatment option to help patients with long COVID cope better and recover quicker from this condition.

Participants will wear a nasal canula (placed in their nostrils) to inhale a gas from a machine that they will be trained to use at home. In one 3-week period, the machine will deliver hydroxy gas (treatment) and in a separate 3-week period the machine will deliver normal air (placebo). The order of the treatment or placebo periods will be randomized and separated by a minimum of 3-weeks during which the participants will not use the machine ('washout' period). Neither the participant nor the investigators will know which 3-week period is the treatment and which is the placebo phase. Participants will visit the laboratory (or be tested at home) at the start and end of each 3-week period.

Testing will involve measuring physical ability (handgrip strength, how far they can walk in 6 minutes, how many times they can stand up and sit down in a minute), breathing problems (how hard they can blow out, how breathless they feel), cognitive ability (how quickly they can mark out a trail based on numbers and letters), and state of mind (mood).

The investigators hypothesize that compared to inhaling placebo, inhaling the hydroxy gas will produce greater improvement in physical ability, relieve breathing problems, and enhance cognitive ability and mood, thereby showing that it can relieve key symptoms of long COVID

ELIGIBILITY:
Inclusion Criteria:

* Any moderate or severe pain, breathlessness, or fatigue associated with long COVID
* live within an hour's drive of the Oxford Brookes campus

Exclusion Criteria:

* Pre-existing secondary diseases; tumors, mental health conditions, chronic respiratory conditions such as Chronic Obstructive Pulmonary Disease (COPD), and cardiac disease
* Previous requirement of ICU treatment due to COVID
* Acute or chronic infections or no pre-existing autoimmune diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Breathlessness | Week 0 and Week 4 (just before and after the first 3 week period of home-administration), Week 6 and week 10 (just before and after the start of the second 3 week period of home-administration).
  Total dyspnoea score in the preceding 2 weeks, quantified from the D-12 questionnaire (% maximum score). Sample size estimate was based on this measure.

SECONDARY OUTCOMES:
Exertional dyspnea | Week 0 and Week 4 (just before and after the first 3 week period of home-administration), Week 6 and week 10 (just before and after the start of the second 3 week period of home-administration)
  Change in total dyspnoea score from rest to peak exercise quantified using the D12 questionnaire
Physical capacity (muscle fatigue) | Week 0 and Week 4 (just before and after the first 3 week period of home-administration), Week 6 and week 10 (just before and after the start of the second 3 week period of home-administration)
  (i) Distance walked at their own pace during the 6-minute walk test and the number of sit to stands achieved in 1 minute.
  (ii) Handgrip strength measured using a hand dynamometer as the maximum squeeze (kg) sustained for 5 second (iii) Peak expiratory flow rate (PEF) achieved by blowing into a Wright's peak flow meter as hard as possible (Liters per minute)
Psychological state and cognitive ability | Week 0 and Week 4 (just before and after the first 3 week period of home-administration), Week 6 and week 10 (just before and after the start of the second 3 week period of home-administration)
  (i) Mood cluster scores for "sedation", "discontentment", and "tension" derived from the Bond Lader mood questionnaire (%full scale) (ii) Time taken to complete a trail marking task based on joining sequential numbers and/or letters
General long COVID symptom burden | Week 0 and Week 4 (just before and after the first 3 week period of home-administration), Week 6 and week 10 (just before and after the start of the second 3 week period of home-administration)
  Overall % score on the long COVID Symptom Burden Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shakeeb H Moosavi, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No